CLINICAL TRIAL: NCT04394091
Title: Post-treatment Ultrasensitive Positron Emission Tomography in Nasopharyngeal Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Chief Physician, Sun Yat-sen University
Other Study IDs: ultrasensitive PET/CT in NPC
Record Dates: First submitted 2020-05-12; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: high-sensitivity PET CT; PET CT
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PET CT and ultrasensitive PET CT: Patients receiving chemoradiotherapy will receive a dedicated FDG PET/CT and ultrasensitive PET CT protocol 12 weeks after the end of IMRT .
  Interventions: Device: ultrasensitive PET CT

INTERVENTIONS:
Device: ultrasensitive PET CT — A 194-cm-long total-body positron emission tomography/computed tomography (PET/CT) scanner (uEXPLORER), has been constructed to offer a transformative platform for human radiotracer imaging in clinical research and healthcare. Its total-body coverage and exceptional sensitivity provide opportunities for innovative studies of physiology, biochemistry, and pharmacology.
  Other Names: PET CT

SUMMARY:
NPC Patients receiving IMRT treatment will receive a dedicated FDG PET/CT and high-sensitivity PET/CT protocol simultaneously in the follow-up of Locally Advanced Nasopharyngeal Carcinoma. Hence we establish this prospective cohort study.

DETAILED DESCRIPTION:
Newly-diagnosed patients with stage III or IV non-metastatic Nasopharyngeal Carcinoma (AJCC 8th) will be recruited. All subjects receiving chemoradiotherapy will undergo a baseline integrated [18F]fluoro-2-deoxy-D-glucose (FDG) positron emission tomography/computed tomography (PET/CT) scan or traditional follow-up examination before the start of chemoradiotherapy.

NPC Patients receiving IMRT treatment will receive a dedicated FDG PET/CT and high-sensitivity PET/CT protocol simultaneously 12 weeks after the end of chemoradiotherapy (primary endpoint).

The results of FDG PET/CT and high-sensitivity PET/CT analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be informed of the investigational nature of this study and given written informed consent.
* Aged between 18-70, male/female.
* Staged III or IV (AJCC 8th) NPC patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma (including differentiated type and undifferentiated type, WHO II and III).
* Received induction chemotherapy and/or concurrent chemoradiotherapy. ECOG scale 0-1.
* Fertile women should practice contraception during the study period.
* HGB ≥90g/L ,WBC ≥4*109/L , PLT ≥100*109/L,
* With normal liver function test (ALT and AST ≤2.5*ULN, TBil ≤2.0*ULN)
* With normal renal function test (serum creatinine ≤1.5*ULN)

Exclusion Criteria:

* Women in pregnancy or lactation
* Prior malignancy except adequately treated basal cell, squamous cell skin cancer, or cervical cancer in situ.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.
* Already involved in other clinical trial.
* Mental disorder, civil disability, limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NPC patients after induction chemotherapy and concurrent chemoradiotherapy or concurrent chemoradiotherapy alone
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
results of ultrasensitive and normal PET CT | 6 months
  The results of the two tests were compared to verify the specificity and sensitivity of ultrasensitive PET CT in post treatment NPC

CONTACTS AND LOCATIONS:
Overall Officials: Haiqiang Mai, Dr, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang X, Cherry SR, Xie Z, Shi H, Badawi RD, Qi J. Subsecond total-body imaging using ultrasensitive positron emission tomography. Proc Natl Acad Sci U S A. 2020 Feb 4;117(5):2265-2267. doi: 10.1073/pnas.1917379117. Epub 2020 Jan 21. PMID 31964808
- [Result] Zhang X, Xie Z, Berg E, Judenhofer MS, Liu W, Xu T, Ding Y, Lv Y, Dong Y, Deng Z, Tang S, Shi H, Hu P, Chen S, Bao J, Li H, Zhou J, Wang G, Cherry SR, Badawi RD, Qi J. Total-Body Dynamic Reconstruction and Parametric Imaging on the uEXPLORER. J Nucl Med. 2020 Feb;61(2):285-291. doi: 10.2967/jnumed.119.230565. Epub 2019 Jul 13. PMID 31302637
- [Result] Lv Y, Lv X, Liu W, Judenhofer MS, Zwingenberger A, Wisner E, Berg E, McKenney S, Leung E, Spencer BA, Cherry SR, Badawi RD. Mini EXPLORER II: a prototype high-sensitivity PET/CT scanner for companion animal whole body and human brain scanning. Phys Med Biol. 2019 Mar 21;64(7):075004. doi: 10.1088/1361-6560/aafc6c. PMID 30620929